CLINICAL TRIAL: NCT00800046
Title: A Study of Percutaneous Repair of Functional Mitral Regurgitation Using the Ancora Heart, Inc. AccuCinch® Ventricular Repair System - The CINCH-2 Study
Acronym: CINCH-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1436
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Mitral Regurgitation; Mitral Valve Regurgitation; Functional Mitral Regurgitation
Keywords: Mitral valve; Mitral regurgitation; Functional mitral regurgitation; MR; FMR; Heart valve; Mitral valve insufficiency; Valve repair; Valve disorder; Cardiac surgery
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- AccuCinch® Ventriculoplasty System (Experimental): Patients meeting the enrollment criteria will be treated with the AccuCinch® Ventriculoplasty System.
  Interventions: Device: AccuCinch® Ventriculoplasty System

INTERVENTIONS:
Device: AccuCinch® Ventriculoplasty System — Mitral valve repair due to functional disease

SUMMARY:
Prospective single-arm study of the AccuCinch® Ventriculoplasty System in the treatment of mitral valve regurgitation through subvalvular mitral repair.

Purpose: To demonstrate the safety, feasibility and potential efficacy of using the AccuCinch® Ventriculoplasty System to reduce mitral valve regurgitation through subvalvular mitral repair.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severity of FMR: ≥ Moderate (i.e., 2+)
* Ejection Fraction: ≥ 20% to ≤60%
* Symptom Status: NYHA II-IVa
* Treatment and compliance with optimal guideline directed medical therapy for heart failure for at least 1 month
* Surgical risk: Subject is eligible for cardiac surgery (specific EuroSCORE (LES or ESII), STS, or comorbidities should demonstrate high risk features)
* Completion of all qualifying diagnostic and functional tests and agrees to comply with study follow-up schedule

Exclusion Criteria:

* Significant organic mitral valve pathology (e.g. myxomatous degeneration, mitral valve prolapse or flail leaflets)
* Myocardial infarction or any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days
* Prior surgical, transcatheter, or percutaneous mitral valve intervention
* Untreated clinically significant coronary artery disease (CAD) requiring revasularization
* Hemodynamic instability: Hypotension (systolic pressure <90 mmHg) or requirement for inotropic support or mechanical hemodynamic support
* Any planned cardiac surgery within the next 6 months (including right heart procedures)
* NYHA class (i.e., non-ambulatory) or ACC/AHA Stage D heart failure
* Fixed pulmonary artery systolic pressure >70 mmHg
* Severe tricuspid regurgitation (per ASE guidelines and graded by the Echo Core Lab)
* Modified Rankin Scale ≥ 4 disability
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
* Mitral valve area less than 4.0 cm2
* Anatomical pathology/contraints preventing appropriate access/ implant of the AccuCinch System
* Renal insufficiency (i.e., eGFR of <30ml/min/1.73m2 ; Stage 4 or 5 CKD)
* Moderate or severe aortic valve stenosis or regurgitation or aortic valve prosthesis Fluoroscopic or echocardiographic evidence of severe aortic arch calcification, mobile aortic atheroma, intracardiac mass, thrombus or vegetation
* Active bacterial endocarditis
* History of stroke within the prior 3 months
* Subjects in whom anticoagulation or antiplatelet therapy is contraindicated
* Known allergy to nitinol, polyester, or polyethylene
* Any prior true anaphylactic reaction to contrast agents; defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure.
* Life expectancy < 1 year due to non-cardiac conditions
* Currently participating in another interventional investigational study
* Implant or revision of any rhythm management device (CRT or CRTD) or implantable cardioverter defibrillator within 1 month
* Absence of CRT with class I indication criteria for biventricular pacing (left bundle branch block pattern and QRS duration ≥150 ms)
* On high dose steroids or immunosuppressant therapy
* Female subjects who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Safety through 30 days and reduction in MR acutely and at 30 days. | 30 days

SECONDARY OUTCOMES:
Safety and reduction in MR at 1 year. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Schofer, Prof. Dr., Principal Investigator — Medical Care Center Prof. Mathey, Prof. Schofer, GmbH; Patrick Perier, MD, Principal Investigator — Cardiovascular Center Bad Neustadt
Locations (8):
- Medical University of Vienna, Vienna, Austria
- Germany (6):
  - University Hospital Freiburg-Bad Krozingen, Bad Krozingen
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau
  - St.-Johannes-Hospital, Dortmund
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Cardiovascular Center Frankfurt, Frankfurt
  - Medical Care Center Hamburg University Cardiovascular Center, Hamburg
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania